CLINICAL TRIAL: NCT03537612
Title: Sensorial and Physiological Mechanism-based Assessments of Perioperative Pain
Acronym: RCT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Do to our inability to meet recruitment targets - Sponsor stopped funding. Looking for new sponsor and protocol modifications
Sponsor: Dr. Jean A. Ouellet, MD, FRCSC (Other)
Responsible Party: Sponsor-Investigator, Dr. Jean A. Ouellet, MD, FRCSC, Deputy Chief of Staff, Shriners Hospitals for Children
Organization: Shriners Hospitals for Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN1701
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Scoliosis
Keywords: Post-operative pain
MeSH Terms: conditions — Scoliosis; Pain, Postoperative | interventions — Clonidine; Morphine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Opt-Clonidine (Experimental): Intrathecal Clonidine 1 mcg/kg (up to 75 mcg) immediately post-op; Clonidine pill TID Post-op Day 1-5 (liquid version available if subject cannot swallow capsule)
  Interventions: Drug: Clonidine
- Sub-opt-Clonidine (Experimental): Intrathecal Clonidine 1 mcg/kg (up to 75 mcg) immediately post-op; Clonidine pill TID Post-op Day 1-5 (liquid version available if subject cannot swallow capsule)
  Interventions: Drug: Clonidine
- Opt-Morphine (Active Comparator): Intrathecal spinal morphine (5 mcg / kg) immediately post-op; Placebo pill TID Post-op Day 1-5 (liquid version available if subject cannot swallow capsule)
  Interventions: Other: Morphine
- Sub-opt-Morphine (Active Comparator): Intrathecal spinal morphine (5 mcg / kg) immediately post-op; Placebo pill TID Post-op Day 1-5 (liquid version available if subject cannot swallow capsule)
  Interventions: Other: Morphine

INTERVENTIONS:
Drug: Clonidine — Intrathecal Clonidine 1 mcg/kg (up to 75 mcg) immediatey post-op; 100 mcg capsule TID Post op day 1-5 (liquid version available if subject cannot swallow capsule)
  Arms: Opt-Clonidine; Sub-opt-Clonidine
Other: Morphine — Intrathecal spinal morphine (5 mcg / kg) immediatey post-op; Placebo capsule TID Post op day 1-5 (liquid version available if subject cannot swallow capsule)
  Arms: Opt-Morphine; Sub-opt-Morphine

SUMMARY:
The overall goal of this proposal is to determine if quantitative sensory testing (QST) assessing pain modulation can be used as a clinical tool to optimize perioperative pain management. The central hypothesis is that the identification of patient's sensory pain profile allows personalizing therapeutic approaches to improve individualized pain management and thus prevents pain chronicity.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate if pre-operative QST can identify if patients will have high pain intensity peri-operatively and at 6 months post-operatively. Evaluation of the intensity and chronicity of pain and the function of the descending inhibitory system through a short QST procedure before surgery and six months after surgery will be carried out. In addition, evaluation of the patient's physical and emotional functioning, and exploration of the potential biological underlying mechanisms will also be assessed at the same time points.

The secondary objective of this study is to determine if the peri-operative use of an alpha-2 adrenergic receptor agonist enhances the efficacy of the descending inhibitory system of patients with sub-optimal CPM efficacy before surgery by decreasing pain after surgery. Consequently, this pharmacological intervention may also reduce the incidence of acute and chronic pain after surgery. Evaluation of the pain intensity and the function of the descending inhibitory system through a short QST procedure six weeks after surgery and six months after surgery in patients receiving Clonidine or placebo during the perioperative period will be done. In addition, evaluation of the patient's physical and emotional functioning, and exploration the potential biological underlying mechanisms at the same time points will be assessed.

Lastly, evaluation of potential biomechanical alterations in 3D related to pain in children reporting presence of back pain pre and post spine surgery will be looked at.

The hypothesis is that patients undergoing spine surgery with poor inhibitory pain response will have less pain in the immediate and long-term period when treated prophylactically with Clonidine in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Females* aged between 10 and 21 years old
* Scheduled to undergo anterior or posterior spinal fusion surgery for AIS with instrumentation
* Ability to adequately understand and respond to outcome measures
* No previous major orthopedic surgery
* Any ethnic background

Exclusion Criteria:

* Children with history of allergies to Clonidine or it's excipients in either injection or tablet formulation (see respective monograph)
* Children with history of galactose intolerance
* Children with history of myocardial disease, arrhythmias, cerebrovascular disease, Raynaud's/Thromboangiitis obliterans or chronic renal failure diagnosis based on history and physical
* Children taking anti-hypertensive agents (diuretics, vasodilators, beta-blockers, ace-inhibitors)
* History of depression
* Inability of the child to speak English or French
* Diagnosed with developmental delay that would interfere with understanding the questions being asked (autism, mental retardation)
* Children with major chronic medical conditions (ASA status III or higher)
* Pregnancy excluded by an in hospital testing the night before surgery

Ages: 10 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
QST | 6 months
  Evaluate if pre-operative QST can identify if patients will have high pain intensity peri-operatively and at 6 months post-operatively.

SECONDARY OUTCOMES:
Clonidine | 6 months
  Peri-operative use of an alpha-2 adrenergic receptor agonist enhances the efficacy of the descending inhibitory system of patients with sub-optimal CPM efficacy before surgery by decreasing pain after surgery.

OTHER OUTCOMES:
3D Images 3D Biomechanical Alterations | 6 months
  Evaluate the potential biomechanical alterations in 3D related to pain in children reporting presence of back pain pre and post spine surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jean A Ouellet, MD, Principal Investigator — Shriners Hospital for Children - Canada
Locations (1):
- Shriners Hospitals for Children - Canada, Montreal, Quebec, Canada

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT03537612/Prot_SAP_000.pdf